CLINICAL TRIAL: NCT03244813
Title: Evaluation of the Impact of a Personalized Program of Adapted Physical Activates in Patients With Parkinson Disease
Acronym: ACTIPARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NIMAO/2016/EV-01
Record Dates: First submitted 2017-06-16; First posted 2017-08-10 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The medical team assessing patient functional capacities and caregiver burden at 3 and 6 months will not know which treatment the patient received
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted physical activity (Experimental)
  Interventions: Other: Personalized activity program
- Standard care (No Intervention)

INTERVENTIONS:
Other: Personalized activity program — Targeted physical activity
  Arms: Adapted physical activity

SUMMARY:
Our study aims to compare the effects of a standard care plan to one using adapted physical activity in patients with Parkinson Disease. Using actigraphy as an evaluation measure will allow the collection of quantitative and objective data related to activity in contrast to questionnaires which are more subjective and dependent on self-representation. In addition, the evaluation of the caregiver's actigraphy and hardship (Zarit scale) will provide interesting data from this population.

ELIGIBILITY:
Inclusion Criteria:

* The patient and their carer have given their free and informed consent and signed the consent form
* The patient must be insured of the beneficiary of an insurance policy
* The patient is available for the 6 month follow-up
* The patient is between 40 and 80 years old
* The patient has experienced symptoms of Parkinson Disease for at least 5 years and is in a stable state (no medical event or change of treatment in at least 1 month)
* The functional impact and duration of fluctuations is ≥3 (MDS UPDRS)
* The patient can walk autonomously, including using a technical aid
* The patient does not have any regular physical activity excluding physiotherapy sessions
* The patient has daily help from a caregiver

Exclusion Criteria:

* The subject and/or their caregiver is participating in another study
* The subject and/or their caregiver is in a period of exclusion determined by a previous study
* The patients is under judicial protection or state guardianship
* It proves impossible to give the patient and/or the caregiver clear information
* The patients and/or the caregiver reuses to sign the consent form
* The patient is pregnant or breast feeding
* The patient has anxiety or depression (Score HAD≥ 11/14), cardiac or respiratory failure (stress test), vesico-sphincter problems preventing normal practice of a physical activity, a contraindication to adapted physical activities
* The patient cannot walk
* Muscular tremor preventing the actigraphy measurement. Outside normal range values for UPDRS measures of: 3.15) postural tremor of the hands; 3.16) action tremor of the hands; 3.17) amplitude of rest tremor

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the impact of an adapted physical activity (APA) program versus standard care on the activity of patients with Parkinson Disease | 3 months
  previous weeks' activity measured by actigraphy

SECONDARY OUTCOMES:
Activity of patients in both groups | 6 months
  previous weeks' activity measured by actigraphy
Activity of patients in both groups | 6 months
  assessed by international physical activity questionnaire
Quality of life of patients undertaking APA verses standard care | 3 months
  Assessed by PDG-39 questionnaire
Quality of life of patients undertaking APA verses standard care | 6 months
  Assessed by PDG-39 questionnaire
Risk of fall of patients undertaking APA verses standard care | 3 months
  measured by Timed Up and Go test
Risk of fall of patients undertaking APA verses standard care | 6 months
  measured by Timed Up and Go test
Risk of fall of patients undertaking APA verses standard care | 3 months
  measured by Tinetti Falls Efficacy Scale
Risk of fall of patients undertaking APA verses standard care | 6 months
  measured by Tinetti Falls Efficacy Scale
Risk of fall of patients undertaking APA verses standard care | 3 months
  measured by 0-10 scale
Risk of fall of patients undertaking APA verses standard care | 6 months
  measured by 0-10 scale
Endurance and speed of walking of patients undertaking APA verses standard care | 3 months
  6 minute walk test
Endurance and speed of walking of patients undertaking APA verses standard care | 6 months
  6 minute walk test
Activity of the care giver | 3 months
  previous weeks' activity measured by actigraphy
Activity of the care giver | 6 months
  previous weeks' activity measured by actigraphy
Evaluation of the care burden of care giver | 3 months
  Zarit scale
Evaluation of the care burden of care giver | 6 months
  Zarit scale
Grip strength | Day 0
  Pinch test
Grip strength | 6 months
  Pinch test
Patient dependence | Day 0
  Activities of Daily Living
Patient dependence | 6 months
  Activities of Daily Living
Level of dementia at Day | Day 0
  Instrumental Activities of Daily Living
Level of dementia at Day | 6 months
  Instrumental Activities of Daily Living

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886